CLINICAL TRIAL: NCT02430181
Title: An Open-label, Dose-ranging, Proof-of-Concept Study to Evaluate the Safety and Efficacy of Lonafarnib With and Without Ritonavir Boosting in Patients Chronically Infected With Delta Hepatitis (HDV) (LOWR-1)
Brief Title: Lonafarnib With and Without Ritonavir in HDV (LOWR-1)
Acronym: LOWR-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIG-300; Application #1128309 (Other: Turkish Regulatory Authority)
Record Dates: First submitted 2015-04-21; First posted 2015-04-30 (Estimated); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Chronic Hepatitis D Infection
MeSH Terms: interventions — lonafarnib; peginterferon alfa-2a; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- lonafarnib - I (Experimental): lonafarnib 200 mg BID; n=3
  Interventions: Drug: lonafarnib
- lonafarnib - II (Experimental): lonafarnib 300 mg BID; n=3
  Interventions: Drug: lonafarnib
- lonafarnib - III (Experimental): lonafarnib 100 mg TID; n=3
  Interventions: Drug: lonafarnib
- lonafarnib/PEG IFN-a - I (Experimental): lonafarnib 100 mg BID + PEG IFN-a 180 ug QW; n=3
  Interventions: Drug: lonafarnib; Drug: peginterferon alfa-2a
- lonafarnib/PEG IFN-a - II (Experimental): lonafarnib 200 mg BID + PEG IFN-a 180 ug QW; n=3
  Interventions: Drug: lonafarnib; Drug: peginterferon alfa-2a
- lonafarnib/PEG IFN-a - III (Experimental): lonafarnib 300 mg BID + PEG IFN-a 180 ug QW; n=2
  Interventions: Drug: lonafarnib; Drug: peginterferon alfa-2a
- lonafarnib/ritonavir (Experimental): lonafarnib 100 mg BID + ritonavir 100 mg QD; n=3
  Interventions: Drug: lonafarnib; Drug: ritonavir

INTERVENTIONS:
Drug: lonafarnib — antiviral farnesyl transferase inhibitor
  Other Names: Sarasar; EBP994
Drug: peginterferon alfa-2a — immunomodulator
  Other Names: Pegasys; pegylated interferon-alfa; PEG IFN-alfa; PEG IFN-a
  Arms: lonafarnib/PEG IFN-a - I; lonafarnib/PEG IFN-a - II; lonafarnib/PEG IFN-a - III
Drug: ritonavir — CYP 3A4 inhibitor, lonafarnib booster
  Other Names: Norvir; RTV
  Arms: lonafarnib/ritonavir

SUMMARY:
To Evaluate the Safety and Efficacy of Lonafarnib with and without Ritonavir Boosting in Adults With Genotype 1 Chronic Hepatitis D Virus (HDV) Infection (LOWR-1).

DETAILED DESCRIPTION:
Chronic delta hepatitis is a serious form of chronic liver disease caused by infection with the hepatitis D virus (HDV), a small RNA virus that requires farnesylation of its major structural protein (HDV antigen) for replication. Twenty-one subjects with chronic delta hepatitis will be randomized to receive one of seven different doses of lonafarnib. Dosing will occur over 4-12 weeks, depending on treatment arm, and during that time, evidence of antiviral response will be assessed by frequent measurements of HDV-RNA. The primary therapeutic endpoint will be an improvement in quantitative serum HDV RNA levels after treatment with lonafarnib therapy. The primary safety endpoint will be the ability to tolerate the drug at the prescribed dose for the treatment duration. Several secondary endpoints will be measured, including side effects, ALT levels, and symptoms. Therapy will be stopped for intolerance to lonafarnib. This study is designed as a phase 2a study assessing the safety, tolerance and antiviral activity of seven dose combinations of lonafarnib with and without ritonavir boosting.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 65 years of age who are diagnosed with HDV by PCR
* Chronic hepatitis D infection, genotype 1, documented by a positive anti-HDV Ab test at least of 6 months duration and detectable HDV RNA by PCR within 3 months to study entry
* Liver biopsy within the last two years
* Positive viral load by quantitative PCR
* Electrocardiogram (ECG) shows no acute ischemia or clinically significant abnormality and a QT/QTc interval <450 milliseconds - using Bazett's correction
* Females of childbearing potential (intact uterus and within 1 year since the last menstrual period) should be non-lactating and have a negative serum pregnancy test. In addition, these subjects should agree to use one of the following acceptable birth control methods throughout the study:

  1. abstinence
  2. surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) six months minimum
  3. IUD in place for at least six months
  4. barrier methods (condom or diaphragm) with spermicide
  5. surgical sterilization of the partner (vasectomy for six months)
  6. hormonal contraceptives for at least three months prior to the first dose of study drug
* Willing and able to comply with study procedures and provide written informed consent

Exclusion Criteria:

* Participation in a clinical trial with or use of any investigational agent within 30 days of Study Visit 1
* Patients co-infected with HIV
* Patients with screening tests positive for HCV, or anti-HIV Ab
* History of decompensated cirrhosis within the past year
* Active jaundice defined by total bilirubin > 2.0 excluding Gilbert's disease
* INR ≥ 1.5
* Eating disorder or alcohol abuse within the past 2 years, excessive alcohol intake (> 20 g per day for females (1.5 standard alcohol drinks) or > 30 g per day for males (2.0 standard alcohol drinks) (a standard drink contains 14 g of alcohol: 12 oz of beer, 5 oz of wine or 1.5 oz of spirits) (1.0 fluid oz (US) = 29.57 mL).
* Drug abuse within the last six months with the exception of cannabinoids and their derivatives
* Patients with absolute neutrophil count (ANC) < 1500 cells/mm^3; platelet count < 100,000 cells/mm^3; hemoglobin < 12 g/dL for women and < 13 g/dL for men; abnormal TSH,T4, or T3 or thyroid function not adequately controlled; or serum creatinine concentration ≥ 1.5 times upper limit of normal (ULN)
* History or clinical evidence of any of the following:

  1. variceal bleeding, ascites, hepatic encephalopathy, CTP score > 6, decompensated liver disease or any other form of non-viral hepatitis
  2. immunologically mediated disease (e.g., rheumatoid arthritis, inflammatory bowel disease, severe psoriasis, systemic lupus erythematosus) requiring more than intermittent nonsteroidal anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids (inhaled asthma medications are allowed)
  3. any malignancy within 3 years except for basal cell skin cancer
  4. significant or unstable cardiac disease (e.g., angina, congestive heart failure, uncontrolled hypertension, history of arrhythmia)
  5. chronic pulmonary disease (e.g., chronic obstructive pulmonary disease) associated with functional impairment
  6. severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization 2
* Patients with a body mass index > 30 kg/m^2
* Concomitant drugs known to prolong the QT interval

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Yurdaydin, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical School, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Eiger BioPharmaceuticals, Inc. company website — http://eigerbio.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lonafarnib/PEG IFN-a - I: lonafarnib 100 mg BID + PEG IFN-a 180 ug QW; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
- Lonafarnib/PEG IFN-a - II: lonafarnib 200 mg BID + PEG IFN-a 180 ug QW; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
- Lonafarnib/PEG IFN-a - III: lonafarnib 300 mg BID + PEG IFN-a 180 ug QW; n=2
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
Period: Overall Study
Arm/Group | Lonafarnib - I | Lonafarnib - II | Lonafarnib - III | Lonafarnib/PEG IFN-a - I | Lonafarnib/PEG IFN-a - II | Lonafarnib/PEG IFN-a - III | Lonafarnib/Ritonavir
Started | 3 | 3 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Patients aged 18-65 years with documented HBsAg, anti-delta positivity for at least 6 months, and compensated liver disease were eligible after evaluation for other forms of chronic liver disease. Patients were required to have detectable HDV-RNA levels at screening, platelet counts >/= 100,000/mm3, absolute neutrophil count >/= 1,500 /mm3, and international normalized ratio <1.5. Patients with hepatocellular carcinoma were excluded.
Groups:
- Lonafarnib 200 mg BID: lonafarnib 200 mg BID; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
- Lonafarnib 300 mg BID: lonafarnib 300 mg BID; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
- Lonafarnib 100 mg TID: lonafarnib 100 mg TID; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
- 100 mg BID Lonafarnib/PEG IFN-a: lonafarnib 100 mg BID + PEG IFN-a 180 ug QW; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
- 200 mg BID Lonafarnib/PEG IFN-a: lonafarnib 200 mg BID + PEG IFN-a 180 ug QW; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
- 300 mg BID Lonafarnib/PEG IFN-a: lonafarnib 300 mg BID + PEG IFN-a 180 ug QW; n=3
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
- Total: Total of all reporting groups
Arm/Group | Lonafarnib 200 mg BID | Lonafarnib 300 mg BID | Lonafarnib 100 mg TID | 100 mg BID Lonafarnib/PEG IFN-a | 200 mg BID Lonafarnib/PEG IFN-a | 300 mg BID Lonafarnib/PEG IFN-a | Lonafarnib/Ritonavir | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 20
Age, Continuous [Mean (Full Range); unit: years] | 59 [57 to 63] | 40 [36 to 46] | 46 [40 to 51] | 41 [22 to 52] | 46 [35 to 53] | 49 [48 to 49] | 51 [42 to 61] | 49 [22 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 7
  Male | 1 | 2 | 1 | 2 | 3 | 1 | 3 | 13
Region of Enrollment [Number; unit: participants]
  Turkey | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Quantitative Serum HDV RNA Levels After 4-12 Weeks of Lonafarnib-based Therapy
Description: log HDV RNA decline from baseline to end of treatment (4-12 weeks of lonafarnib-based therapy)
Time Frame: 4-12 weeks
Measure: Mean (Full Range); unit: log IU/mL
Groups:
- 300 mg BID Lonafarnib/PEG IFN-a: lonafarnib 300 mg BID + PEG IFN-a 180 ug QW; n=2
  lonafarnib: antiviral farnesyl transferase inhibitor
  PEG IFN-a: immunomodulator
Arm/Group | Lonafarnib 200 mg BID | Lonafarnib 300 mg BID | Lonafarnib 100 mg TID | 100 mg BID Lonafarnib/PEG IFN-a | 200 mg BID Lonafarnib/PEG IFN-a | 300 mg BID Lonafarnib/PEG IFN-a | Lonafarnib/Ritonavir
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 3
log IU/mL | 0.03 [-1.17 to 1.83] | -1.78 [-2.28 to -1.46] | -1.3 [-1.61 to -0.52] | -1.85 [-2.4 to -1.33] | 0 [0 to 0] | 0 [0 to 0] | -1.2 [-1.41 to -0.91]

ADVERSE EVENTS:
Arm/Group | Lonafarnib 200 mg BID | Lonafarnib 300 mg BID | Lonafarnib 100 mg TID | 100 mg BID Lonafarnib/PEG IFN-a | 200 mg BID Lonafarnib/PEG IFN-a | 300 mg BID Lonafarnib/PEG IFN-a | Lonafarnib/Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 0/3 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 0/3 | 0/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lonafarnib 200 mg BID (N=3) | Lonafarnib 300 mg BID (N=3) | Lonafarnib 100 mg TID (N=3) | 100 mg BID Lonafarnib/PEG IFN-a (N=3) | 200 mg BID Lonafarnib/PEG IFN-a (N=3) | 300 mg BID Lonafarnib/PEG IFN-a (N=2) | Lonafarnib/Ritonavir (N=3)
dehydration secondary to vomiting and diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lonafarnib 200 mg BID (N=3) | Lonafarnib 300 mg BID (N=3) | Lonafarnib 100 mg TID (N=3) | 100 mg BID Lonafarnib/PEG IFN-a (N=3) | 200 mg BID Lonafarnib/PEG IFN-a (N=3) | 300 mg BID Lonafarnib/PEG IFN-a (N=2) | Lonafarnib/Ritonavir (N=3)
weight loss (Investigations) | 3 | 3 | 2 | 1 | 0 | 0 | 2
diarrhea (Gastrointestinal disorders) | 3 | 3 | 2 | 3 | 0 | 0 | 3
nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 3 | 0 | 0 | 3
fatigue (General disorders) | 3 | 2 | 2 | 1 | 0 | 0 | 2
vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No